CLINICAL TRIAL: NCT06541054
Title: The Effect of Perioperative Heated Sock Use in Preventing Hypothermia During Total Hip Prosthesis Surgery: A Randomized Controlled Trial
Brief Title: The Effect of Perioperative Heated Sock Use in Preventing Hypothermia During Total Hip Prosthesis Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Seval Ulubay, PhD, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Interventional
Record Dates: First submitted 2022-09-04; First posted 2024-08-07 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Hip Fractures; Hip Injuries
MeSH Terms: conditions — Hip Fractures; Hip Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Body temperature, pulse, arterial blood pressure, SPO2 will be measured and recorded every fifteen minutes in the control group one hour before the operation. The patients in the control group will not be dressed in warm socks and general preparations will be made. During the operation, the patient's body temperature, pulse, arterial blood pressure, SPO2 values will be monitored every fifteen minutes and the total amount of drainage during the operation will be recorded in the same department. Body temperature, pulse, arterial blood pressure, SPO2 values, tremors, and total drainage in the postoperative care unit will be recorded every fifteen minutes. Body temperature, heart rate, arterial blood pressure, SPO2 values will be measured after transferring to the bed and every fifteen minutes for a total of 180 minutes, chills, shivering states, and 24-hour total drainage amount will be recorded in the same section.
- experiment group (Experimental): One hour before the operation,warm socks will be put on the experimental group,body temperature,heart rate,blood pressure,SPO2 will be measured and recorded every fifteen minutes.During the surgery,body temperature,heart rate,blood pressure,SPO2 value, drainage amount will be measured and recorded every fifteen minutes.The patient will be transferred to the postoperative care unit with warm socks and will stay on his feet in the postoperative care unit.Body temperature, heart rate,blood pressure,SPO2 values will be recorded every fifteen minutes.He will be transferred from the postoperative care unit to the clinic with socks.will stay. After transferring to the bed,body temperature,heart rate, arterial blood pressure, SPO2 will be recorded every fifteen minutes for a total of 180minutes.Chills,chills and the total drainage amount for 24hours will be recorded in the same section.
  Interventions: Other: WARM SOCKS

INTERVENTIONS:
Other: WARM SOCKS — One hour before the operation,warm socks will be put on the experimental group,body temperature,heart rate,blood pressure,SPO2 will be measured and recorded every fifteen minutes.During the surgery,body temperature,heart rate,blood pressure,SPO2 value, drainage amount will be measured and recorded every fifteen minutes.The patient will be transferred to the postoperative care unit with warm socks and will stay on his feet in the postoperative care unit.Body temperature, heart rate,blood pressure,SPO2 values will be recorded every fifteen minutes.He will be transferred from the postoperative care unit to the clinic with socks.will stay. After transferring to the bed,body temperature,heart rate, arterial blood pressure, SPO2 will be recorded every fifteen minutes for a total of 180minutes.Chills,chills and the total drainage amount for 24hours will be recorded in the same section.
  Arms: experiment group

SUMMARY:
Warm sock application; It has been proven that wearing battery-operated warm socks on patients in the preoperative period strengthens the central thermoregulation system, maintains core body temperature, controls the shivering response, and ensures the subjective thermal comfort of patients.

DETAILED DESCRIPTION:
Preoperative hypothermia, which is one of the problems frequently experienced by patients, during surgical interventions individual and environmental . It develops as a result of the deterioration of the temperature regulation mechanism due to factors such as exposure of tissues and organs, etc. Body temperature is a vital sign, which is regulated by the hypothalamic thermoregulatory center with physical and chemical systems and accepted within normal limits between 36-37.7°C. Hypothermia is defined by the American Association of Perianesthesia Nurses as 36°C below the central temperature. Body temperature between 34-36°C is classified as mild hypothermia, 32-34°C as moderate hypothermia, and below 32°C as severe hypothermia . Hypothermia, which is defined as a decrease in body temperature below 36°C is common in the preoperative period. is a common problem. A decrease in body temperature below 36 °C one hour before anesthesia and up to 24 hours after anesthesia is defined as "preoperative hypothermia". In general, hypothermia is a complication that can affect the length of hospital stay, wound healing, and patient satisfaction.Total hip replacement is surgery to replace a severely damaged hip with an artificial joint. Total hip replacement is a surgical treatment method applied in advanced ages for degenerative joint disease, rheumatoid arthritis, femoral neck fracture and developmental hip dislocation. The aim of total hip replacement is to relieve hip pain, to regain the diminished function of the joint by increasing the range of motion, and to improve the quality of life . Total hip replacement is also applied to young patients with severely damaged and painful hip joints . Patients at high risk of developing hypothermia under anesthesia; being female, patients with a preoperative body temperature below 36°C, patients undergoing sedation and premedication, patients who will undergo major and moderate surgery, patients with concomitant cardiovascular disease, patients undergoing general anesthesia, those over 70 years of age patients, those with systolic blood pressure above 140 mmHg, those with diseases such as heart disease, hypothyroidism, brain tumor, adrenal insufficiency, chronic kidney failure, diabetes mellitus, except for surgical pathology, those with anemia, those with a body mass index below 25 , trauma and burn patients are at risk for hypothermia . Major (neurosurgery, prosthetic surgery, thoracic surgery, etc.) and long-term (> 2 hours) surgical interventions, opening large body spaces, application of cold fluids, blood and blood products, cold and dry anesthetic gases, excessive irrigation, excessive irrigation loss of fluid and blood, lack of muscle movements in the patient, the patient being naked and immobile, wide body surfaces remaining open, and wet dressings cause hypothermia development during surgical intervention . In addition, the likelihood of hypothermia increases with aging. Total hip replacement surgery, which is frequently performed in the elderly due to rheumatoid arthritis, osteoarthritis, osteoporosis, problems affecting the spinal cord and serious extremity injuries is a major intervention and includes many of the risks mentioned for hypothermia. Nurses have a great responsibility in ensuring and maintaining temperature control in the surgical process. Nurses can reduce the development of hypothermia by using active and passive warming methods to maintain the patient's normal body temperature in the preoperative period . Surgical nurses should evaluate and record the hypothermia risk factors, signs and symptoms before the operation, closely monitor the body temperature of the patients, determine and apply appropriate warming methods according to body temperature. In a study by Grossman, it was determined that patients who used heating method in the postoperative period reached their normal body temperature in a shorter time than patients who were not warmed .The mean body temperature of the patients after two hours of warming before surgery was found to be 36.4°C . Kurşun and Dramalı (2011) determined that the patients who were warmed in the postoperative period reached their normal body temperature in a shorter time than the patients who were not heated. Active and passive warming methods are used in the control of hypothermia in surgical patients. In active heating methods, heat is given to the patient by one or more of the ways of external conduction, radiation, and convection. These; are external and internal heating methods. In the external heating method, the heat is given to the patient's skin with active cutaneous heaters. warm socks; In the pre-operative period, wearing pre-warmeḑ stockings has proven effective in maintaining core body temperature, controlling shivering response, and providing patients' subjective thermal comfort. Pre-warmed stockings are a noninvasive, easy-to-wear, painless, and cost-effective method of preventing heat loss. Allows efficient repositioning of the patient and surgical preparation. It also provides comfort to patients, reduces preoperative anxiety and can be applied without a doctor's prescription . The lack of comprehensive studies examining the effect of preoperative active warming on maintaining body temperature during and after surgery and the possibility of explaining the effect of warm socks on maintaining body temperature, warmeḑ socks; It is seen that it strengthens the central temperature regulation system and ultimately maintains core body temperature and can control the shivering response, thus maintaining subjective thermal comfort. The lack of comprehensive studies examining the effect of preoperative active warming on maintaining body temperature during and after surgery and the fact that patients who experienced. Total hip replacement were in the high risk group for hypothermia formed the basis of this study. In the light of all information, in this study, it was aimed to determine the effectiveness of warm stockings, which is one of the active heating methods in prevention, and to contribute to the literature by drawing attention to the risk of hypothermia in patients experiencing.

ELIGIBILITY:
Inclusion Criteria:

* The duration of surgical intervention is between 2 and 4 hours,
* Ability to read, write, understand and communicate in Turkish,
* Voluntary participation in the study,
* Does not require follow-up in intensive care before or after surgery,
* Dementia, alzheimer etc. absence of disease affecting cognitive functions,
* Absence of a disease that may affect thermoregulation due to systemic effects such as chronic obstructive pulmonary disease (COPD), cancer, intracranial benign/malignant tumor, epilepsy, multiple sclerosis, Parkinson's disease, and thyroid-related diseases,
* Absence of drug use that may affect thermoregulation,
* It is not uncomfortable to wear heat socks during application.

Exclusion Criteria:

* Mental retardation and the presence of any psychiatric disorder,
* Being addicted to alcohol and drugs,
* Dementia, alzheimer etc. have a disease that affects cognitive functions,
* Having drug use that may affect thermoregulation,
* Discomfort from wearing heat socks during application,
* Having any disease that affects tissue perfusion,
* Presence of any peripheral arterial and venous disease,
* The need for intensive care before or after surgery

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
The Effect of Perioperative Heated Sock Use in Preventing Hypothermia During Total Hip Prosthesis Surgery: A Randomized Controlled Trial | 36 weeks
  As a result of the measurement in this study: Body temperature is measured tympanically. Hypothermia is generally classified based on cases where the body temperature falls below 35.0 °C. Hypothermia symptoms may vary as body temperature drops, so hypothermia is divided into three levels according to its severity.Body Temperature: Monitoring body temperature before and after surgery. Specifically, evaluating whether preoperative warm sock application helps maintain body temperature within normal ranges.
  Target Body Temperature: Assessing whether the targeted body temperature range (e.g., 36-37°C) for preventing hypothermia is achieved.

CONTACTS AND LOCATIONS:
Overall Officials: SEVAL ULUBAY, phd, Study Director — IUC
Locations (1):
- Seval Ulubay, Samsun, Atakum/Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
After the approval of the board, warm socks and sensitive scales to be used in my thesis work were provided. Permission was obtained from Samsun Gazi State Hospital, where the research would be conducted. Ethics Committee Approval from Samsun Health Sciences University Samsun Training and Research Hospital and permission from Samsun Health Directorate. Groups were determined by randomization over a pre-calculated sample. It was planned to start the pilot study after randomization and to proceed to the data collection phase of the study by making the necessary corrections after the pilot study. In addition, in this process, the writing of the introduction, general information, materials and methods section of the thesis will begin.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2022-2023
Access Criteria: sevalulubay@gmail.com

REFERENCES:
- [Result] Lauronen SL, Kalliomaki ML, Aho AJ, Kalliovalkama J, Riikonen JM, Makinen MT, Leppikangas HM, Yli-Hankala AM. Thermal suit in preventing unintentional intraoperative hypothermia during general anaesthesia: a randomized controlled trial. Acta Anaesthesiol Scand. 2017 Oct;61(9):1133-1141. doi: 10.1111/aas.12945. Epub 2017 Jul 25. PMID 28741744

DOCUMENTS (3):
  • Study Protocol (2022-12-31): https://cdn.clinicaltrials.gov/large-docs/54/NCT06541054/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-31): https://cdn.clinicaltrials.gov/large-docs/54/NCT06541054/SAP_001.pdf
  • Informed Consent Form (2022-12-31): https://cdn.clinicaltrials.gov/large-docs/54/NCT06541054/ICF_002.pdf